CLINICAL TRIAL: NCT03866044
Title: Unravelling the Alteration of Brain Structure and Function in Parkinson´s Disease With Ultra-high Field MRI
Acronym: 7TPD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Danish Research Centre for Magnetic Resonance (Other)
Collaborators: Bispebjerg Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: H-18021857
Record Dates: First submitted 2019-02-07; First posted 2019-03-07 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parkinson's Disease (PD): Patients with Parkinson's Disease meeting the following criteria:
  Inclusion criteria:
  * Aged 18 or more.
  * Clinically established or probable PD according to the MDS Clinical Diagnostic Criteria for Parkinson's Disease
  * Signed informed consent
  Exclusion criteria:
  * Pregnancy or breastfeeding
  * History of other neurologic or psychiatric disease
  * Pacemaker or other implanted electronic devices
  * Claustrophobia
- Healthy participants: Healthy participants age- and sex-matched to the PD group.
  Inclusion criteria:
  * Age- and sex-matched to PD group (aged 18 or more)
  * Signed informed consent
  Exclusion criteria:
  * Pregnancy or breastfeeding
  * History of neurologic or psychiatric disease
  * Pacemaker or other implanted electronic devices
  * Claustrophobia

SUMMARY:
Parkinson's Disease (PD) is a neurodegenerative disease characterized by a range of disabling motor- and non-motor symptoms caused by a loss of neurons in neuromodulatory brainstem nuclei. Typical motor symptoms include bradykinesia, rigidity and tremor. Non-motor symptoms are diverse and include REM sleep behaviour disorder, hyposmia, autonomic dysfunction, depression, apathy and cognitive impairment. The motor symptoms can in some degree be attributed to degeneration of the substantia nigra (SN) and a deficiency of dopamine (DA) availability, and DA replacement therapy can partially alleviate motor symptoms. The role of nigral degeneration on non-motor symptoms is however less clear. In addition to nigral degeneration, the noradrenergic (NA) locus coeruleus (LC) also undergoes severe degeneration in PD. Again, it is unclear how LC degeneration contributes to motor and non-motor symptoms.

Ultra-high resolution structural magnetic resonance imaging (MRI) provides the opportunity to assess alterations of the affected nuclei in detail and functional MRI (fMRI) can map activation in the neuronal populations as a measure of DA and NA function.

DETAILED DESCRIPTION:
BACKGROUND Parkinson's disease (PD) is a multi-system neurodegenerative disease affecting a subset of vulnerable cells in various brain structures, including brain stem nuclei. Selective degeneration of dopamine (DA) producing neurons in the pars compacta of the substantia nigra (SNc) is a key neuropathological feature in PD and gives rise to the classical motor symptoms which can be symptomatically treated by dopamine replacement therapy. Yet the link between DA and PD extends far beyond the motor system, pertaining to core aspects of cognition that are supported by dopamine signalling: For instance, there is converging evidence that reward computations and motivational drive are significantly affected by PD and its dopaminergic treatment. Noradrenaline (NA) producing cells of the pontine nucleus locus coeruleus (LC) are also affected in PD with early and severe degeneration. Although the LC is the main source of NA in the brain, and NA has been shown to be an important neuromodulator, it is unclear how neurodegeneration of the LC contributes to motor and non-motor symptoms in PD.

PD and the dopaminergic system Several midbrain nuclei contain cell groups that synthesize the neurotransmitter DA and project from the ventral tegmental area (VTA) and SNc to cortical areas and the striatum. It has recently been suggested that VTA and SNc have distinct roles in reinforcement learning: dopamine bursts from VTA are thought to reinforce stimulus values, while the SNc is specifically important for action values. Since PD preferentially affects the ventral tier of the SNc leading to the motor symptoms, it has been hypothesized that dopaminergic treatment leads to an "overdosing" of the less impaired pathways from VTA to striatum.

PD and the noradrenergic system Parallel to the degeneration of dopaminergic neurons in SNc, noradrenergic neurons in the pontine locus coeruleus (LC) exhibit Lewy pathology and undergo a marked degeneration early on in PD which exceeds that of dopaminergic SNc neurons. The LC is the largest source of noradrenaline (NA) to the brain, and exerts neuromodulatory effects through extensive ascending projections to the entire cerebral cortex. The loss of NA neuromodulation associated with PD might contribute to both motor and non-motor symptoms and could potentially be a therapeutic target, however the effect and significance of NA deficiency in PD pathogenesis is to date not fully understood. The LC is thought to be involved in the modulation of attention and arousal and also in the processing of emotion. The role of LC neurodegeneration and the resulting decrease in noradrenaline levels to the pathophysiology of PD is not fully understood. However, a large number of studies in humans and animals support a double role of noradrenergic cell loss in PD; a contribution to motor- and non-motor symptoms as well as a facilitation of DA neurodegeneration.

AIMS The overall purpose of the study is to map structural and functional changes in the subcortical dopaminergic and noradrenergic networks that mediate cognition, attention and emotion in PD.

The study aims to:

* Measure PD related neurodegeneration on 7T sMRI in ROIs corresponding to neuromodulatory brainstem nuclei: Substantia nigra pars compacta, nigrosome-1, ventral tegmental area & locus coeruleus
* Predict disease severity by multivariate pattern of neurodegeneration measures in these areas.
* Map the relationship between the autonomic arousal response to arousing stimuli, neural activity in the noradrenergic arousal network and the degree of neurodegeneration in noradrenergic brain regions.
* Investigate the effects of neurodegeneration in the core dopaminergic nuclei (SNc and VTA) and dopaminergic medication on the midbrain striatal network mediating action-value and stimulus-value learning.

HYPOTHESES

Structural changes of SN and LC integrity:

1. Participants with PD will have significantly decreased signal on MTw-imaging in the SN and LC quantified as reduced contrast ratios in SN/cerebral peduncle and LC/pontine tegmentum.
2. SN and LC volumes, calculated as the sum of supra-threshold voxels in the regions of SN and LC, will be significantly decreased in participants with PD.
3. Accelerated iron accumulation in SN and nigrosome-1 will lead to an increased hypointensity of the SN and a loss of a distinct nigrosome-1 region on SWI, R2* and QSM.
4. R2* and QSM values in SN on Quantitative Susceptibility Mapping will be significantly higher in participants with PD.
5. Motor impairment (UPDRS-3 subscore) can be predicted by multivariate pattern analysis of MTw- and SWI-images of the SN.
6. Measures of LC structural integrity will correlate with non-motor symptoms, specifically apathy and depression.

   Functional changes:
7. Participants with PD will have significantly decreased functional activation in a region corresponding to the LC when exposed to arousing stimuli.
8. Functional activation in the LC will correlate with LC structural integrity.
9. Autonomic arousal responses (pupil response and skin conductance response) will correlate with LC structural integrity and functional activation.
10. In healthy controls, there will be increased SN-dorsal striatal connectivity for action value learning, increased VTA-ventral striatal connectivity for stimulus value learning.
11. In PD patients off their medication, there will be reduced SN-dorsal striatal connectivity. This will impair action value learning while stimulus value learning will only be mildly affected.
12. Dopaminergic medication restores dopamine levels in the dorsal striatum and "overdoses" ventral striatum. Medication will restore (at least partially) SN-dorsal striatal connectivity and dorsal striatal activity which will lead to largely unimpaired action value learning. "Overdosing" will result in exaggerated VTA-ventral striatal connectivity and exaggerated ventral striatal activity. In subjects with strong ventral striatal "overdosing" inappropriate stimulus value learning might occur.

RESEARCH PLAN Part 1: 7T and 3T structural MRI to map structural changes in SN and LC and their clinical correlates in PD.

Participants: 60 patients with idiopathic PD (aged 18 or more), 20 age-matched healthy control subjects.

Ultra-high field MRI. All participants will be scanned using a research-only 7T Achieva MR System (Philips, Best, The Netherlands) located at Hvidovre Hospital. MR-scanning will be performed with a dual transmit, 32-channel receive head coil (Nova Medical Products), including a neuromelanin sensitive, magnetization transfer weighted (MTw) sequence at 0.4x0.4x1.0mm resolution, a susceptibility weighted imaging (SWI) sequence at 0.4mm isotropic resolution and a multi-echo quantitative R2* sequence at 1.0mm isotropic resolution. Additionally, all participants will be scanned using a 3T Siemens Prisma MR system.

Additional examinations: Outside the scanner, motor and non-motor symptoms (UPDRS, Unified Parkinson's Disease Rating Scale & NMSS, Non-Motor Symptom Scale), cognition (MoCA, Montreal Cognitive Assessment), apathy (LARS, Lille Apathy Rating Scale), depression (BDI-II, Beck's Depression Inventory), impulse control disorders (QUIP, Parkinson's Disease Impulsive-Compulsive Disorders Questionnaire), impulsivity (BIS-11, Barratt Impulsiveness Scale), and handedness (EHI, Edinburgh Handedness Inventory) will be assessed.

Part 2: 7T fMRI to assess DA and NA dysfunction in PD Participants: A sub-group of individuals who participated in part 1 will be asked to participate in Part 2: It is expected that 20 patients and all the healthy participants are able to lie sufficiently still to cooperate in a fMRI experiment.

Participants will be scanned again with the 7T Achieva MR system using a reduced transverse field-of-view covering the SN and LC. Structural imaging will include a 1.0 mm isotropic T1w sequence for co-registration. High-spatial resolution functional Blood Oxygen Level Dependent (BOLD) (fMRI) will be used to map the functional activations of SN and LC in two task-fMRI paradigms. For the assessment of NA activation, a paradigm utilizing auditory stimuli and visual stimuli with arousing content (IAPS, International Affective Picture System) will be administered in two separate sessions; first inside the scanner, and secondly outside the scanner, during which autonomic responses to the stimuli (pupil responses and skin conductance responses) are recorded. In the second paradigm, participants will be gambling on a virtual slot machine with two handle bars in two different colours where one of the handles can be pushed, the other pulled. Participants have MRI-compatible joysticks to pull or push the handles of the virtual slot machine. Depending on the block, the action performed (pulling or pushing the handles, irrespective of their colour) or the stimulus colour (yellow or blue, irrespective of whether they can be pushed or pulled) are predictive of reward and punishment (one option has a higher reward probability than the other, these have to be learnt via feedback). Reward probabilities are changing repeatedly and unannounced.

Patients will undergo the experiments twice on two separate days, on and off PD medication, in a randomized, balanced order. Healthy participants will also undergo the experiments on two separate days.

ELIGIBILITY:
1. Parkinson's Disease (PD) group

   Inclusion criteria:
   * Aged 18 or more.
   * Clinically established or probable PD according to the Movement Disorder Society Clinical Diagnostic Criteria for Parkinson's Disease
   * Signed informed consent

   Exclusion criteria:
   * Pregnancy or breastfeeding
   * History of other neurologic or psychiatric disease
   * Pacemaker or other implanted electronic devices
   * Claustrophobia
2. Healthy participants age- and sex-matched to the PD group:

Inclusion criteria:

* Age- and sex-matched to PD group (aged 18 or more)
* Signed informed consent

Exclusion criteria:

* Pregnancy or breastfeeding
* History of neurologic or psychiatric disease
* Pacemaker or other implanted electronic devices
* Claustrophobia

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the ambulatory care at the Department of Neurology, Bispebjerg Hospital and through private practicing neurologists. As part of the clinical assessment relevant patients with PD will be asked if they would be interested in participating in the study. Also, letters with invitation to participate in the study will be sent to patients with PD in treatment at the clinics. Participants will also be recruited from the general population via advertisements.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2018-09-19 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
SN contrast ratio on neuromelanin sensitive images | Baseline
  Mean SI(SN)/mean SI(cerebral peduncles), SI=signal intensity. We expect that PD patients will have decreased SN contrast ratio compared with age-matched healthy participants and that SN contrast ratio will correlate with UPDRS-3 subscore.
SN volume on neuromelanin sensitive images | Baseline
  Voxels in SN with mean SI > SI+2 standard deviations(cerebral peduncles) , SI=signal intensity).
  We expect that PD patients will have decreased SN volume compared with age-matched healthy participants and that SN volume will correlate with UPDRS-3 subscore.
LC contrast ratio on neuromelanin sensitive images | Baseline
  Mean SI(LC)/mean SI(pontine tegmentum), SI=signal intensity. We expect that PD patients will have decreased LC contrast ratio compared with age-matched healthy participants and that LC contrast ratio will correlate with NMSS, LARS and BDI-II scores.
LC volume on neuromelanin sensitive images | Baseline
  Voxels in LC with mean SI > SI+4 standard deviations(pontine tegmentum), SI=signal intensity).
  We expect that PD patients will have decreased LC volume compared with age-matched healthy participants and that LC volume will correlate with NMSS, LARS and BDI-II scores.
Total SN iron accumulation: SWI | Baseline
  SN mean signal intensity on SWI. We expect that PD patients will have lower mean SN SWI signal intensity compared to healthy.
Total SN iron accumulation: R2* | Baseline
  SN mean R2* values (unit=1/s). We expect that PD patients will have higher mean SN R2* values compared to healthy.
Total SN iron accumulation: QSM | Baseline
  SN mean QSM values (unit=ppb). We expect that PD patients will have higher mean SN QSM values compared to healthy.
Nigrosome-1 iron accumulation: SWI | Baseline
  Nigrosome-1 signal visibility on SWI assessed by blinded raters. We expect that iron accumulation in nigrosome-1 will be greater in PD patients leading to a loss of discrimination on SWI.
Nigrosome-1 iron accumulation: R2* | Baseline
  Mean R2* values in the nigrosome-1 region (unit=1/s). We expect that PD patients will have higher R2* values in the nigrosome-1 region.
Nigrosome-1 iron accumulation: QSM | Baseline
  Mean QSM values in the nigrosome-1 region (unit=ppb). We expect that PD patients will have higher QSM values in the nigrosome-1 region.
Functional brain activation pattern in the LC, SN, VTA, and striatum | ON & OFF PD medication in a period within 24 weeks from baseline.
  Revealed by task related blood oxygenation level dependent (BOLD) signal changes.
  We expect that functional activation in these regions will be attenuated in PD patients corresponding to their loss of brainstem nuclei integrity (see hypotheses).
Motor disease severity | Baseline
  Unified Parkinson's Disease Rating Scale (UPDRS)-3 subscore (Motor severity, range 0-108, higher values = worse outcome). Measured while subjects are taking their usual medication.
Overall disease severity | Baseline
  Total Unified Parkinson's Disease Rating Scale (UPDRS) score (sum of all 4 subscores listed below, range 0-199, higher values = worse outcome), UPDRS-1 (Cognitive and mental disease severity, range 0-16, higher values = worse outcome), UPDRS-2 (disease severity in relation to activities of daily living, range 0-52, higher values = worse outcome) and UPDRS-3 (Motor severity, range 0-108, higher values = worse outcome), UPDRS-4 (Complications of therapy, range 0-23, higher values = worse outcome) subscores. Measured while subjects are taking their usual medication.
Non-motor disease severity | Baseline
  Total Non-Motor Symptom Scale (NMSS) score (range 0-360, higher values = worse outcome). Measured while subjects are taking their usual medication.
Modified Hoehn and Yahr Staging | Baseline
  Modified Hoehn and Yahr Staging (Crude measure of disease severity, range 0-5, higher score = worse outcome). Measured while subjects are taking their usual medication.
Schwab and England Activities of Daily Living Scale | Baseline
  Schwab and England Activities of Daily Living Scale (Measure of ADL function, range 100-0%, higher score = better outcome). Measured while subjects are taking their usual medication.
Apathy | Baseline
  Total Lille Apathy Rating Scale (LARS) score (range -36-36, higher score = better outcome).
Mood | Baseline
  Total Beck's Depression Inventory-II (BDI-II) score (range 0-63, lower score = better outcome).
Autonomic emotional-arousal response: Pupillary response | ON & OFF PD medication in a period within 24 weeks from baseline.
  Change in pupil size in response to arousing stimuli compared with non-arousing stimuli (unit=difference in mm).
  We expect that PD patients will have a smaller pupillary response following arousing stimuli compared to healthy participants.
Autonomic emotional-arousal response: Skin conductance response | ON & OFF PD medication in a period within 24 weeks from baseline.
  Change in skin conductance (unit=micro Siemens) in response to arousing stimuli compared with non-arousing stimuli.
  We expect that PD patients will show an attenuated skin conductance response to arousing stimuli compared to healthy participants.
Behavioural outcome measures: Choices | ON & OFF PD medication in a period within 24 weeks from baseline.
  Learning in reinforcement learning paradigm: Choices, reaction times, parameters describing degree of action-value vs. stimulus value learning from computational model.
Behavioural outcome measures: Reaction times | ON & OFF PD medication in a period within 24 weeks from baseline.
  Learning in reinforcement learning paradigm: Reaction times (unit=ms) describing degree of action-value vs. stimulus value learning from computational model.
Behavioural outcome measures: Model parameters | ON & OFF PD medication in a period within 24 weeks from baseline.
  Learning in reinforcement learning paradigm: Model parameters describing degree of action-value vs. stimulus value learning from computational model.

CONTACTS AND LOCATIONS:
Overall Officials: Hartwig R Siebner, DMSci, Principal Investigator — Danish Research Centre for Magnetic Resonance
Locations (2):
- Denmark (2):
  - Department of Neurology, Copenhagen University Hospital Bispebjerg, Copenhagen
  - Danish Research Centre For Magnetic Resonance, Copenhagen University Hospital Hvidovre, Hvidovre

IPD SHARING:
Plan to Share IPD: Undecided